CLINICAL TRIAL: NCT00064129
Title: A Phase I Study of Repetitive Dosing of Anti-CTLA-4 Antibody (Ipilimumab) in Combination With GM-CSF in Patients With Metastatic, Androgen-Independent Prostate Cancer
Brief Title: Ipilimumab and Sargramostim in Treating Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00036; NCI-2009-00036 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCSF-02558; CDR0000309054; NCI-6032; 02558 (Other: UCSF Medical Center-Mount Zion); 6032 (Other: CTEP); NCT01648361 (obsolete NCT alias)
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Recurrent Prostate Carcinoma; Stage IV Prostate Cancer AJCC v7
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ipilimumab; CTLA-4 Antigen; sargramostim; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (monoclonal antibody, colony-stimulating factors) (Experimental): Patients receive ipilimumab IV over 90 minutes on day 1 and sargramostim (GM-CSF) SC on days 1-14. Treatment repeats every 28 days for 4-6 courses. GM-CSF continues beyond 4 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of ipilimumab until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Some patients undergo blood sample collection periodically for laboratory and pharmacokinetic studies. Samples are analyzed for human anti-human antibodies, IgG antibodies to ipilimumab semi-quantitative ELISA assay, and plasma concentrations of ipilimumab via quantitative ELISA assay.
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Biological: Sargramostim

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Biological: Sargramostim — Given SC
  Other Names: 23-L-Leucinecolony-Stimulating Factor 2; DRG-0012; Leukine; Prokine; rhu GM-CFS; Sagramostim; Sargramostatin

SUMMARY:
This phase I trial is studying the side effects and best dose of ipilimumab when given with sargramostim in treating patients with metastatic prostate cancer. Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Colony-stimulating factors, such as sargramostim, may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (MDX-010) (ipilimumab) administered with sargramostim (GM-CSF) in patients with metastatic androgen-independent prostate cancer. (Phase I) II. Determine the safety of this regimen in these patients. (Phase I) III. Evaluate the efficacy as measured by reduction in PSA associated with combining GM-CSF with CTLA-4 blockade with ipilimumab at a dosage of 3 mg/kg given monthly x 6 doses (d1 of courses 1-6). (Cohort Expansion)

SECONDARY OBJECTIVES:

I. Determine the T-cell immunity and T-cell response in patients treated with this regimen. (Phase I) II. Determine the pharmacokinetics of MDX-010 in these patients. (Phase I) III. Determine the prostate-specific antigen and/or objective responses in patients treated with this regimen. (Phase I) IV. Determine the percentages of activated, naive, and memory T-cells. (Cohort Expansion) V. Determine the measurement of T-cell response to describe epitopes from prostate antigens including PSA, PSMA, and PAP. (Cohort Expansion) VI. Quantitate T-cell response to antigens in patients with relevant HLA allele using HLA*0201 tetramers. (Cohort Expansion) VII. Evaluate the toxicity of this regimen in these patients. (Cohort Expansion) VIII. Determine the initial efficacy as measured by reduction in PSA associated with combining GM-CSF with CTLA-4 blockade with ipilimumab at a dosage of 3 mg/kg given monthly x 6 doses (d1 of courses 1-6). (Cohort Expansion) IX. Determine objective response by post-therapy measurable disease changes using RECIST criteria. (Cohort Expansion)

OUTLINE: This is a multicenter, dose-escalation study of ipilimumab.

Patients receive ipilimumab intravenously (IV) over 90 minutes on day 1 and sargramostim (GM-CSF) subcutaneously (SC) on days 1-14. Treatment repeats every 28 days for 4-6 courses. GM-CSF continues beyond 4 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of ipilimumab until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Some patients undergo blood sample collection periodically for laboratory and pharmacokinetic studies. Samples are analyzed for human anti-human antibodies, IgG antibodies to ipilimumab semi-quantitative ELISA assay, and plasma concentrations of ipilimumab via quantitative ELISA assay.

Patients are followed at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer

  * Metastatic disease
* Progressive disease after prior androgen deprivation as defined by at least 1 of the following criteria:

  * Patients with measurable disease must have an increase of at least 20% in the sum of the longest diameter of target lesions OR the appearance of 1 or more new lesions
  * Patients with nonmeasurable disease must have a positive bone scan and a prostate-specific antigen (PSA) level of at least 5 ng/mL, which has risen on at least 2 successive occasions at least 2 weeks apart*

    * At least 1 PSA level must be obtained at least 4 weeks after flutamide (6 weeks after bicalutamide or nilutamide)
* Testosterone no greater than 50 ng/dL

  * Patients with no prior orchiectomy must continue luteinizing hormone-releasing hormone agonist therapy
* No history or radiologic evidence of CNS metastases
* Performance status - ECOG 0-2
* At least 12 weeks
* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8 g/dL
* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT and SGPT no greater than 2.5 times ULN
* Creatinine no greater than 1.5 times ULN
* No significant cardiovascular disease
* No New York Heart Association class III or IV congestive heart failure
* No active angina pectoris
* No myocardial infarction within the past 6 months
* Not pregnant or nursing
* Fertile patients must use effective contraception prior to, during, and for 3 months after study participation
* No history of autoimmune disease including, but not limited to, any of the following:

  * Autoimmune hemolytic anemia
  * Ulcerative and hemorrhagic colitis
  * Endocrine disorders (e.g., thyroiditis, hyperthyroidism, hypothyroidism of immune etiology, autoimmune hypophysitis/hypopituitarism, or adrenal insufficiency)
  * Sarcoid granuloma
  * Myasthenia gravis
  * Polymyositis
  * Guillain-Barre syndrome
  * Systemic lupus erythematosus
  * Rheumatoid arthritis
  * Inflammatory bowel disease
* No other medical or psychiatric illness that would preclude study participation or giving informed consent
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or stage I or II cancer currently in complete remission
* No prior immunotherapy (e.g., vaccines or investigational)
* No other concurrent colony-stimulating factors
* No prior chemotherapy
* No concurrent chemotherapy
* See Disease Characteristics
* At least 4 weeks since prior systemic corticosteroids
* At least 4 weeks since other prior hormonal therapy, including megestrol and finasteride
* No concurrent systemic steroid therapy except inhaled or topical steroids
* No other concurrent hormonal therapy

  * Hormones administered for nondisease-related conditions (e.g., insulin for diabetes) allowed
* At least 4 weeks since prior radiotherapy and recovered
* More than 8 weeks since prior radiopharmaceuticals (e.g., strontium chloride Sr 89 and samarium Sm 153 lexidronam pentasodium)
* Prior irradiation of a symptomatic lesion or one that may produce disability (e.g., unstable femur) allowed
* No concurrent palliative radiotherapy
* See Disease Characteristics
* At least 4 weeks since prior herbal products known to decrease PSA levels (e.g., PC-SPES or saw palmetto)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2003-05-13 (Actual); Primary Completion 2011-01-10 (Actual); Study Completion 2012-10-01 (Actual)

PRIMARY OUTCOMES:
MTD of the combination of ipilimumab with GM-CSF that results in < 33% DLT | Continuously
  Graded according to the National Cancer Institute (NCI) common toxicity criteria, version 3.0. Results will be tabulated by dose cohort and overall for this trial. DLT is defined by any of the following that are attributable to therapy: any >= grade 4 toxicity, any ocular toxicity considered immune mediated and requiring systemic steroids, any grade 3 toxicity considered immune mediated that cannot be controlled with systemic steroids.

SECONDARY OUTCOMES:
Adaptive immunity | Baseline, days 1 and 14 of courses 1 and 2, day 1 of courses 3-6, and then day 1 of every other course throughout treatment
  Measured through peripheral blood collection. Three and four-color immunofluorescence and flow cytometric analysis will be employed to determine relative numbers of activated T cells. Specifically, percentages of T cells (CD3+, CD4+ or CD8+) expressing the activation markers HLA-DR, CD25 and CD69 will be determined. Also, percentages of naive (CD45RA+) and memory (CD45RO+) T cells will be determined.
PSA and/or objective response for measurable disease | Day 1
  Evaluated according to Response Evaluation Criteria in Solid Tumors (RESIST) criteria. PSA Response will be evaluated according to the recommendations from National Cancer Institute PSA Working Group. 95% confidence interval will be provided.
Safety of the regimen | Continuously
  Graded according to the NCI common toxicity criteria, version 3.0.
Anti-idiotype antibody (human anti-human antibodies [HAHA]) development | Baseline, before each ipilimumab infusion and 2 months after the last infusion of antibody
  A semi-quantitative ELISA assay will be used to detect IgG antibodies to Ipilimumab in the plasma samples.
Pharmacokinetic (PK) Studies | Prior to and 60 minutes after all infusions, and at 1 and 2 months after the last ipilimumab infusion
  Determined using a quantitative ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Small, Principal Investigator — UCSF Medical Center-Mount Zion
Locations (1):
- UCSF Medical Center-Mount Zion, San Francisco, California, United States

REFERENCES:
- [Derived] Cham J, Zhang L, Kwek S, Paciorek A, He T, Fong G, Oh DY, Fong L. Combination immunotherapy induces distinct T-cell repertoire responses when administered to patients with different malignancies. J Immunother Cancer. 2020 May;8(1):e000368. doi: 10.1136/jitc-2019-000368. PMID 32376721
- [Derived] Kavanagh B, O'Brien S, Lee D, Hou Y, Weinberg V, Rini B, Allison JP, Small EJ, Fong L. CTLA4 blockade expands FoxP3+ regulatory and activated effector CD4+ T cells in a dose-dependent fashion. Blood. 2008 Aug 15;112(4):1175-83. doi: 10.1182/blood-2007-11-125435. Epub 2008 Jun 3. PMID 18523152